CLINICAL TRIAL: NCT06562296
Title: Multicenter, Prospective, Randomized Controlled Matriarch Trial Evaluating Several Cellular, Acellular, and Matrix-like Products (CAMPs) and Standard of Care Versus SOC Alone of Nonhealing Diabetic Foot and Venous Leg Ulcers
Brief Title: Study Evaluating Several CAMPs in Nonhealing Diabetic Foot and Venous Leg Ulcers
Acronym: CAMPLIFE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cellution Biologics (Industry)
Collaborators: SerenaGroup, Inc. (Network); LifeCell (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CELLBIO-2024-001
Record Dates: First submitted 2024-08-12; First posted 2024-08-20 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Foot Ulcer; Venous Leg Ulcer
Keywords: diabetic foot ulcer; venous leg ulcer; DFU; VLU; ulcer
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer; Ulcer | interventions — cancer procoagulant; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- AIC for DFUs (Experimental): Participants with a diabetic foot ulcer (DFU) will receive treatment with an Amnion-Intermediate-Chorion sheet product, a dehydrated multilayer human placental tissue derived from donated human tissue, and weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Interventions: Other: Amnion-Intermediate-Chorion; Procedure: Standard of Care
- AIC for VLUs (Experimental): Participants with a venous leg ulcer (VLU) will receive treatment with an Amnion-Intermediate-Chorion sheet, a dehydrated multilayer human placental product derived from donated human tissue, and weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Interventions: Other: Amnion-Intermediate-Chorion; Procedure: Standard of Care
- ACA for DFUs (Experimental): Participants with a diabetic foot ulcer (DFU) will receive treatment with an Amnion-Chorion-Amnion sheet allograft product, a dehydrated trilayer human placental tissue derived from donated human tissue, and weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Interventions: Other: Amnion-Chorion-Amnion; Procedure: Standard of Care
- ACA for VLUs (Experimental): Participants with a venous leg ulcer (VLU) will receive treatment with an Amnion-Chorion-Amnion allograft sheet, a dehydrated trilayer human placental product derived from donated human tissue, and weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Interventions: Other: Amnion-Chorion-Amnion; Procedure: Standard of Care
- Standard of Care (Active Comparator): Beginning at the screening visit, participants will receive weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Other: Amnion-Intermediate-Chorion — Dehydrated human placental multilayer allograft from derived donated human tissue. AIC contains amnion and chorion layers as well as basement membrane and trophoblast.
  Other Names: AIC
  Arms: AIC for DFUs; AIC for VLUs
Other: Amnion-Chorion-Amnion — Dehydrated human placental trilayer allograft derived from donated human tissue.
  Other Names: ACA
  Arms: ACA for DFUs; ACA for VLUs
Procedure: Standard of Care — Standard of care is to establish a clean, healthy wound bed and optimize the wound environment to have the best chance of healing the wound. This is achieved through wound cleansing, debridement, offloading and moisture balance.
  Other Names: SOC

SUMMARY:
The purpose of this study is to determine how well multiple CAMPs (Cellular, Acellular and Matrix-Like Products) and Standard of Care work when compared to Standard of Care alone in achieving complete closure of diabetic foot and venous leg ulcers.

DETAILED DESCRIPTION:
Chronic wounds affect a significant percentage of patients over their lifetime. For example, diabetic foot ulcers (DFU) are a major health complication that affect up to 15% of individuals with diabetes mellitus over their lifetime. The treatment of chronic wounds is extremely challenging as ulcers such as DFUs and Venous Leg Ulcers (VLUs) may not respond to standard of care (SOC) treatment and frequently become infected.

Advanced wound products like CAMPs have become an important strategy in the treatment of these chronic wounds by trapping and binding the patients' own cells to rebuild the dermis layer of the skin to aid in healing.

This study will evaluate the clinical utility of Multiple CAMPs in the closure of diabetic foot ulcers and venous leg ulcers in subjects in comparison to Standard of Care treatment.

ELIGIBILITY:
Inclusion Criteria for DFU:

Potential subjects are required to meet all the following criteria for enrollment into the study and subsequent randomization.

* Subjects must be at least 18 years of age or older.
* Subjects must have a diagnosis of type 1 or 2 Diabetes mellitus.
* At randomization subjects must have a target ulcer with a minimum surface area of 0.7 cm2 and a maximum surface area of 5.0 cm2 measured post debridement.
* The target ulcer must have been present for a minimum of 4 weeks and a maximum of 52 weeks of standard of care prior to the initial screening visit.
* The target ulcer must be located on the foot with at least 50% of the ulcer below the malleolus.
* The target ulcer must be Wagner 1 or 2 grade, extending at least through the dermis or subcutaneous tissue and may involve the muscle provided it is below the medial aspect of the malleolus. The ulcer may not include exposed tendon or bone.
* The affected limb must have adequate perfusion confirmed by vascular assessment. Any of the following methods performed within 3 months of the first screening visit are acceptable:

  1. ABI ≥ 0.7 and ≤ 1.3;
  2. TBI ≥ 0.6;
  3. TCOM ≥ 40 mmHg;
  4. PVR: biphasic.
* If the subject has two or more ulcers, they must be separated by at least 2 cm. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
* The subject must consent to using the prescribed off-loading method for the duration of the study.
* The subject must agree to attend the weekly study visits required by the protocol.
* The subject must be willing and able to participate in the informed consent process.

Exclusion Criteria for DFU:

Potential subjects meeting any of the following criteria will be excluded from enrollment and subsequent randomization.

* A subject known to have a life expectancy of < 6 months is excluded.
* The subject is excluded if the target ulcer is not secondary to diabetes.
* If the target ulcer is infected or if there is cellulitis in the surrounding skin.
* If there is evidence of osteomyelitis complicating the target ulcer.
* Subject cannot have an infection in the target ulcer or in a remote location that requires systemic antibiotic therapy.
* A subject receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of Prednisone per day or equivalent) or cytotoxic chemotherapy is excluded.
* The topical application of steroids to the ulcer surface within one month of initial screening is not permitted.
* A subject with a previous partial amputation on the affected foot is excluded if the resulting deformity impedes proper offloading of the target ulcer.
* The subject is excluded if the surface area of the target ulcer has reduced in size by more than 20% in the 2 weeks prior to the initial screening visit ("historical" run-in period).

Photographic planimetry is not required for measurements taken during the historical run-in period (e.g. calculating surface area using length x width is acceptable).

* The subject is excluded if the surface area measurement of the Target ulcer decreases by 20% or more during the 2-week screening phase: the 2 weeks from the initial screening visit (S1) to the TV-1/randomization visit, during which time the subject received SOC.
* A subject is excluded if they are malnourished: a score of less than 17 on the Mini Nutritional Assessment (MNA).
* A Subject with an acute Charcot foot, or an inactive Charcot foot, that impedes proper offloading of the target ulcer is excluded.
* Women who are pregnant or considering becoming pregnant within the next 6 months are excluded.
* A subject with end stage renal disease requiring dialysis is excluded.
* A subject who, in the opinion of the investigator, has a medical or psychological condition that may interfere with study assessments is excluded.
* A subject treated with hyperbaric oxygen therapy or a Cellular Acellular, or Matrix-like Product (CAMP) in the 30 days prior to the initial screening visit is excluded.
* A subject with a known sensitivity to ofloxacin, vancomycin, or amphotericin antibiotics is excluded.
* Participation in a clinical trial involving treatment with an investigational product within the previous 30 days.

Inclusion Criteria for VLU:

Potential subjects are required to meet all the following criteria for enrollment in the study.

* Subjects must be at least 21 years of age or older.
* At randomization subjects must have a target ulcer with a minimum surface area of 1 cm2 and a maximum surface area of 20 cm2 measured post-debridement.
* The target ulcer must have been present for a minimum of 4 weeks and a maximum of 52 weeks of standard of care prior to the initial screening visit.
* No visible signs of healing objectively, less than 40% reduction in wound size in the last 4 weeks.
* The affected limb must have adequate perfusion confirmed by vascular assessment. Any of the following methods performed within 3 months of the first screening visit are acceptable:

  1. ABI between 0.7 and ≤ 1.3;
  2. TBI ≥ 0.6;
  3. TCOM ≥ 40 mmHg;
  4. PVR: biphasic.
* If the potential subject has two or more ulcers, they must be separated by at least 2 cm post-debridement. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
* The potential subject must agree to attend the weekly study visits required by the protocol.
* The potential subject must be willing and able to participate in the informed consent process.

Exclusion Criteria for VLU:

Potential subjects meeting any of the following criteria will be excluded from enrollment in the study.

* The potential subject is known to have a life expectancy of < 6 months.
* The target ulcer is infected, requires systemic antibiotic therapy, or there is cellulitis in the surrounding skin.
* The target ulcer exposes tendon or bone.
* There is evidence of osteomyelitis complicating the target ulcer.
* The potential subject is receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of prednisone per day or equivalent) or cytotoxic chemotherapy or is taking medications that the PI believes will interfere with wound healing (e.g., biologics).
* The potential subject has applied topical steroids to the ulcer surface within one month of initial screening.
* The potential subject has glycated hemoglobin (HbA1c) greater than or equal to 12% within 3 months of the initial screening visit.
* The surface area of the target ulcer has reduced in size by more than 20% in the 2 weeks prior to the initial screening visit ("historical" run-in period). MolecuLight Imaging Device is not required for measurements taken during the historical run-in period (e.g., calculating surface area using length X width is acceptable).
* The surface area measurement of the target ulcer decreases by 20% or more during the active 2-week screening phase: the 2 weeks from the initial screening visit (SV-1) to the TV-1 visit during which time the potential subject received SOC.
* Women who are pregnant or considering becoming pregnant within the next 6 months.
* The potential subject has end stage renal disease requiring dialysis.
* Participation in a clinical trial involving treatment with an investigational product within the previous 30 days.
* A potential subject who, in the opinion of the investigator, has a medical or psychological condition that may interfere with study assessments.
* The potential subject was treated with hyperbaric oxygen therapy (HBOT) or a Cellular, Acellular, Matrix-like Product (CAMP) in the 30 days prior to the initial screening visit.
* The subject has a malnutrition indicator score <17 as measured on the Mini Nutritional Assessment.
* A subject has a wound with active or latent infection is excluded.
* A subject with a disorder that would create unacceptable risk of post-operative complications is excluded.
* A subject with a known sensitivity to ofloxacin, vancomycin, or amphotericin antibiotics is excluded.

Ages: 18 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Percentage of ulcers with complete wound closure | 1-12 weeks
  The percentage of DFU and VLU target ulcers achieving complete wound closure. Closure is defined by 100% re-epithelialization of the ulcer surface without detectable exudate.

SECONDARY OUTCOMES:
Time to complete closure for ulcer | 1-12 weeks
  Time to closure will be determined for each treatment group and compared to Standard Of Care. Closure is defined by 100% re-epithelialization of the ulcer surface without detectable exudate.
Percentage of wound area change for target ulcer | 1-12 weeks
  Percentage wound area changes from week 1 to week 12 will be calculated weekly from measurements with digital photographic planimetry and physical examination.
Incidence of Adverse events | 1-12 weeks
  The incidence of adverse events will be evaluated weekly from the first study visit to wound healing and/or final visit.
Changes to pain associated with the target ulcer | 1-12 weeks
  Change in pain in the target ulcer assessed using the Visual Analog Scale (VAS) from week 1 to week 12. VAS is a tool that uses a 0-10 (no to extreme pain) point scale to measure pain intensity.
Determine changes in Quality of Life | 1-12 weeks
  Changes in quality of life using both the Wound Quality of Life (wQOL) and Forgotten Wound Score (FWS) questionnaires that measure the health-related quality of life (HRQoL) of patients with chronic wounds.
  wQOL questionnaire is scored using a 5-point Likert scale, where 0 means "not at all" and 4 means "very much". Higher scores indicate greater impairment of quality of life. Higher the score indicates lower quality of life. [Time Frame: Visits 1, 4, 8, and 12/Final Visit].
  FWS questionnaire measures 12 activities scored 0-4. Responses are summed and divided by the number of completed items. The mean value is then multiplied by 25 to obtain the total score of 0-100. Higher the score indicates lower quality of life. [Time Frame: Visits 1, 4, 8, and 12/Final Visit].

OTHER OUTCOMES:
Changing in bacterial load | 1-12 weeks
  Changes in chronic inhibitory bacterial load (CIBL) measured using fluorescence imaging [Time Frame: Visits 1, 4, 8, and 12/Final Visit].
Changes in ambulation | 1-12 weeks
  Changes in functional ambulation based on Functional Ambulatory
  Category Scale (FACS) - VLU subjects only. The FACS is a 6-point (0-5) functional walking test that evaluates ambulation ability. Scoring:
  0 indicates that the patient is a non-functional ambulator (cannot walk)
  1, 2 or 3 denotes a dependent ambulator who requires assistance from another person in the form of continuous manual contact (1), continuous or intermittent manual contact (2), or verbal supervision/guarding (3)
  4 or 5 describes an independent ambulator who can walk freely on: level surfaces only (4) or any surface (5=maximum score)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Symphony Research, Jacksonville, Florida
  - Sure Step Foot & Ankle, Cincinnati, Ohio
  - RGV Wound Care Group, Weslaco, Texas
  - Family Foot & Ankle, Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: No